CLINICAL TRIAL: NCT06322927
Title: PatIent exPeRiences and prEFerence of trEatment foR Multiple Myeloma
Acronym: iPREFER
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: CellCentric Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CFTsp231; 24_CPCR_38 (Other: ChristieNHS)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Patient Experience; Treatment Preference; Qualitative Study; Patient Interviews
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Interviews: Participants will be asked to take part in a 30-60 minute interview to understand their treatment preferences. Members of the research team will conduct this either in the clinic or over the phone, as per patient preference.
  Interventions: Other: Patient Interview

INTERVENTIONS:
Other: Patient Interview — Participants will be asked to take part in a 30-60 minute interview to understand their treatment experiences and preferences.

SUMMARY:
This is a qualitative (interview) study to explore the experiences of people receiving treatment for MM and to understand what matters most to participants when making treatment decisions.

DETAILED DESCRIPTION:
People can receive many lines of treatment for multiple myeloma. The investigators would like to understand more about the experiences of people being treated for multiple myeloma including what matters most to participants when considering treatment options, how participants experiences have differed with different treatments and if participants have any treatment preferences. Patients at The Christie who have received five or more lines of treatment for Multiple Myeloma will be eligible to take part in this study. Participants will be asked to take part in an interview which should take approximately 30 minutes to an hour. During the interview, participants will be asked questions regarding their experiences and preference for treatment. Interviews will be conducted either in person or over the phone depending on patient preference. The interviews will be recorded by the research team using a Dictaphone and transcribed by an external transcription service called 1st Class Secretarial. The transcripts of all participant interviews will be reviewed by members of the research team and experiences will be identified and described.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with confirmed MM (per standard disease specific diagnostic criteria)
2. Participants must have received ≥ 5 lines of treatment for MM and fit into one of the below treatment categories:

   1. Subset 1- Participants must have received an oral anti-cancer therapy and a bi-specific antibody treatment.
   2. Subset 2- Participants must have received an oral anti-cancer therapy and if they have not had a bi-specific antibody treatment, they must have received at least one IV therapy.
3. Aged 18 years of age or over
4. Able to provide informed consent
5. Able to communicate in English

Exclusion Criteria:

1. Aged under 18
2. Unable to understand and communicate in the English language
3. Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma who have received at least five lines of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Experience and Preference | 30-60 minutes
  The interview will explore the experiences of people receiving treatment for multiple myeloma and understand what matters most to them when making treatment decisions.

SECONDARY OUTCOMES:
Treatment and Preference Differences | 30-60 minutes
  The interview will explore how experiences have differed across different lines of treatment and determine if people with multiple myeloma have any preferences for particular treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Taylor, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No